CLINICAL TRIAL: NCT02208583
Title: Exploratory Study of Molecular Phenotype Changes and Personalized Treatment for Patients With Castration Resistant Prostate Cancer
Brief Title: Molecular Phenotype Changes and Personalized Treatment for CRPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: E2014064
Record Dates: First submitted 2014-07-29; First posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-06

CONDITIONS: Hormone Refractory Prostate Cancer
Keywords: Molecular phenotypic；CRPC; personalized treatment
MeSH Terms: interventions — Docetaxel; Prednisone; PE regimen; Cisplatin; Etoposide; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AR dependent CRPC (Active Comparator): Assignment to Treatment Group based on druggable gene mutations analysis:
  CRPC patients without druggable gene mutations: Docetaxel & Prednisone; CRPC patients with druggable gene mutations: DP & Targeted drugs
  Interventions: Drug: Docetaxel & Prednisone; Drug: DP & Targeted drugs
- AR independent CRPC (Active Comparator): Assignment to Treatment Group based on druggable gene mutations analysis:
  CRPC patients without druggable gene mutations: cisplatin & Etoposide; CRPC patients with druggable gene mutations: EP & Targeted drugs
  Interventions: Drug: cisplatin & Etoposide; Drug: EP & Targeted drugs

INTERVENTIONS:
Drug: Docetaxel & Prednisone — Docetaxel & Prednisone: Docetaxel 75mg/m2，d1;Prednisone 5mg，bid，d1-21
  Other Names: Taxotere
  Arms: AR dependent CRPC
Drug: DP & Targeted drugs — Docetaxel 75mg/m2，d1; Prednisone 5mg，bid，d1-21;Targeted drugs for PO. Participants with EGFR gene mutation will receive a drug called Gefitinib; Participants with BRAF gene mutations will receive a drug called Vemurafenib; Participants with AKT1 gene mutations will receive a drug called Celecoxib; Participants who have ERBB2 gene mutation will receive a drug called lapatinib; Participants with PDGFRA gene mutations will receive a drug called sunitinib; Participants with PIK3CA gene mutations will receive a drug called Everolimus
  Other Names: Targeted drugs for PO
  Arms: AR dependent CRPC
Drug: cisplatin & Etoposide — cisplatin & Etoposide:cisplatin 25mg/m2，d1-3; Etoposide 100 mg/m2，d1-3
  Other Names: cisplatin and Etoposide for injection
  Arms: AR independent CRPC
Drug: EP & Targeted drugs — cisplatin 25mg/m2，d1-3; Etoposide 100 mg/m2，d1-3; Targeted drugs for po. Participants with EGFR gene mutation will receive a drug called Gefitinib; Participants with BRAF gene mutations will receive a drug called Vemurafenib; Participants with AKT1 gene mutations will receive a drug called Celecoxib; Participants who have ERBB2 gene mutation will receive a drug called lapatinib; Participants with PDGFRA gene mutations will receive a drug called sunitinib; Participants with PIK3CA gene mutations will receive a drug called Everolimus
  Other Names: Targeted drugs for po
  Arms: AR independent CRPC

SUMMARY:
To explore the molecular phenotypic changes and personalized treatment in castration-resistant prostate cancer.

DETAILED DESCRIPTION:
This is a multi-center study to explore the molecular phenotypic changes in castration-resistant prostate cancer by histopathological,immunohistochemical and molecular analysis of cancer related genes in castration-resistant prostate cancer.After patient eligibility is determined, tumor tissue will be acquired from archival or transurethral resection or from re-biopsy specimens from patients with recurrence, visceral metastasis, bone metastases. According to the molecular phenotypic changes, personalized treatment were performed.

Participants will be screened with a full medical history and physical examination, blood and urine tests, and tumor imaging studies. The tumor specimens at diagnosis of prostate cancer should be needed for all the participants.

After assessing for the prostate specific antigen (PSA) level and the tumor molecular phenotypic features,participants will be separated into different treatment groups:

1. Participants with "AR dependent" CRPC (generally with high PSA level and/or high AR expression) and with druggable gene mutations will receive Docetaxel/prednisone+Target drugs.
2. Participants with "AR dependent" CRPC (generally with high PSA level and/or high AR expression) and without druggable gene mutations will receive Docetaxel/ Prednisone.
3. Participants with "AR independent" CRPC (generally without AR expression and/or rapid progression with low PSA level) and with druggable gene mutations will receive Cisplatin/Etoposide+Target drugs.
4. Participants with "AR independent" CRPC (generally without AR expression and/or rapid progression with low PSA level) and without druggable gene mutations will receive Cisplatin/Etoposide.

Participants with druggable gene mutations will receive the corresponding molecular targeted drugs.

Participants with epidermal growth factor receptor (EGFR) gene mutation will receive a drug called Gefitinib, which inhibits a protein called EGFR that is thought to be a key factor in the development and progression of some cancers.

Participants with B-type Raf kinase (BRAF) gene mutations will receive a drug called Vemurafenib, which inhibits a protein called mitogen-activated or extracellular signal-regulated protein kinase kinase (MEK) that is thought to be a key factor in the development and progression of some cancers.

Participants with v-akt murine thymoma viral oncogene homologue 1 (AKT1) gene mutations will receive a drug called Celecoxib, which inhibits a protein called v-akt murine thymoma viral oncogene homologue (AKT) that is thought to be a key factor in the development and progression of some cancers.

Participants who have erythroblastic leukemia viral oncogene homolog 2 (ERBB2) gene mutation will receive a drug called lapatinib, which inhibits some proteins that are thought to be key factors in the development and progression of some cancers.

Participants with PDGFRA gene mutations will receive a drug called sunitinib, which inhibits some proteins that are thought to be key factors in the development and progression of some cancers.

Participants with PIK3CA gene mutations will receive a drug called Everolimus, which inhibits a protein called AKT that is thought to be a key factor in the development and progression of some cancers.

ELIGIBILITY:
Inclusion Criteria:

1. 18 Years and older;
2. patients with CRPC according to European Association of Urology diagnostic criteria ;
3. vital organs functions including bone marrow, heart, liver, kidney are normal;
4. complete pathological specimens including newly diagnosed with prostate cancer and disease progress to CRPC: ① biopsies or surgical specimens (tissue bank or wax block preserved specimens) at diagnosis ; ② re-biopsy specimens,transurethral prostatectomy (TURP) specimens, metastases palliative surgical specimens (tissue bank or wax block preserved specimens) after progress to CRPC; ③ amount sufficient sample for DNA extraction and quality control by up to standard (a) Sample type: None RNA degradation and pollution-free DNA samples; (b) the amount of the sample (single): ≥ 250ng (using agilent liquid platform); (c) sample concentration: ≥ 50 ng / μl (using agilent liquid platform); (d) sample purity: OD 260/280 = 1.8 ~ 2.0 );
5. Then we perform following tests when patients meet the above criteria: ①Histological analysis: Hematoxylin-eosin(HE) staining ②immunohistochemistry(IHC) staining ③ 48 carcinomas associated exon sequencing
6. After performing the above test, enter treatment group ① Docetaxel & Prednisone(DP) : with high PSA and no gene mutation; ② DP + targeted drugs: with high PSA and gene mutations; ③ cisplatin & Etoposide(EP) : low PSA and no gene mutation; ④ EP + targeted drug: Low PSA and gene mutations.
7. All patients enrolled in draw peripheral blood samples 7.5ml and detect circulating tumor cells (CTC) , monitoring efficacy.

8. Willing and able to comply with the program during the study period. 9 before entering clinical trials to provide written informed consent form, and the patient has to know you can withdraw from the study at any time in the study, and without any loss.

10. Agrees to provide blood and tissue specimens. 11 expected survival of> 6 months 12.Karnofsky performance status (KPS)> 60; Eastern Cooperative Oncology Group(ECOG) score 0-2 13 signed informed consent form

Exclusion Criteria:

1. other cancers
2. cognitive inability and mental abnormalities
3. other serious disease or condition

   * severe, uncontrolled internal medicine and infectious diseases
   * severe digestive disorder can not control
   * severe electrolyte imbalance
   * active disseminated intravascular coagulation
   * major organ failure, such as decompensated heart, lung, liver, kidney failure
   * peripheral neuropathy symptoms, NCI grade> Ⅱ degree
4. can not tolerate chemotherapy or refuse chemotherapy
5. using the other test drug or participate other clinical trials
6. can not oral drugs
7. receiving chemotherapy, biological therapy, or other anti-cancer medicine intervals less than 4 weeks
8. Researchers believe patients unsuitable (compliance, we should not follow-up)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Molecular phenotypic changes after acquired resistance of hormonal therapy | 24 months
  The acquired resistance criteria is based on the european criteria for castration resistant prostate cancer.The molecular phenotypic changes including the following observations:1.histopathologic analysis for rebiopsy pathology in CRPC;2.Immunohistochemical staining for androgen receptor(AR),Ki-67,cluster of differentiation 56(CD56),Syn,P53, AURKA,N-myc,retinoblastoma susceptibility(RB), E-cadherin, vimentin;3.Targeting exom sequencing by TruSeq Amplicon Cancer Panel(TSACP) including the hotspot mutation for 48 cancer related genes.
clinical progression free survival(cPFS) | 24months
  cPFS is defined as the time from the start of treatment to disease progression.

SECONDARY OUTCOMES:
Overall Survival(OS) | 24 months
  OS is defined as the time the time from the start of treatment to death.
The relationship between molecular phenotypic changes and OS | 24 months
  The relationship between molecular phenotypic changes and OS means how the molecular phenotypic changes affects OS.

CONTACTS AND LOCATIONS:
Overall Officials: Wang HaiTao, Ph.D, Principal Investigator — Department of Interventional Oncology, Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Department of Interventional Oncology, Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China